CLINICAL TRIAL: NCT00257166
Title: Four Week, Double-Blind, Placebo Controlled Phase III Trial Evaluating The Efficacy, Safety And Pharmacokinetics Of Flexible Doses Of Oral Ziprasidone In Children And Adolescents With Bipolar I Disorder (Manic Or Mixed)
Brief Title: Safety and Efficacy of Ziprasidone in Children and Adolescents With Bipolar I Disorder (Manic or Mixed)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281132
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ziprasidone oral capsules (Experimental)
  Interventions: Drug: Ziprasidone oral capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo oral capsules

INTERVENTIONS:
Drug: Ziprasidone oral capsules — Oral ziprasidone capsules of 20 mg, 40 mg, 60 mg, and 80 mg strength administered BID.
  Arms: Ziprasidone oral capsules
Drug: placebo oral capsules — Oral placebo capsules of 20 mg, 40 mg, 60 mg, and 80 mg strength administered BID.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if flexibly-dosed ziprasidone is safe and effective for the treatment of children and adolescents (ages 10-17) with bipolar I disorder (manic or mixed).

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for Bipolar I disorder (manic or mixed); age 10 - 17 years

Exclusion Criteria:

* Imminent risk of suicide or homicide, as judged by the site investigator; any history of serious or unstable medical illness, including risk for QT prolongation

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (44):
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Altamonte Springs, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Tavares, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Des Plaines, Illinois
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Owensboro, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Pikesville, Maryland
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Clinton Township, Michigan
  - Pfizer Investigational Site, Meridian, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, West Allis, Wisconsin

REFERENCES:
- [Derived] Findling RL, Cavus I, Pappadopulos E, Vanderburg DG, Schwartz JH, Gundapaneni BK, DelBello MP. Efficacy, long-term safety, and tolerability of ziprasidone in children and adolescents with bipolar disorder. J Child Adolesc Psychopharmacol. 2013 Oct;23(8):545-57. doi: 10.1089/cap.2012.0029. Epub 2013 Oct 10. PMID 24111980
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281132&StudyName=Safety%20and%20efficacy%20of%20ziprasidone%20in%20children%20and%20adolescents%20with%20Bipolar%20I%20Disorder%20%28manic%20or%20mixed%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Ziprasidone: Ziprasidone capsule administered orally in 2 divided doses daily in the morning and evening with a starting dose of ziprasidone 20 milligram per day (mg/day) as an evening dose on Day 1. This was followed by dose escalation of 20 mg/day every other day up to a target dose of ziprasidone 120 to 160 mg/day for participants with greater than or equal to [>=] 45 kilogram [kg] weight and ziprasidone 60 to 80 mg/day for participants with less than [<] 45 kg weight over 2 weeks, as per investigator's discretion. Flexible dosing of ziprasidone capsule 80 to 160 mg/day for participants with >= 45 kg weight and ziprasidone capsule 40 to 80 mg/day for participants with <45 kg weight orally in 2 divided doses daily in the morning and evening up to Week 4, as per investigator's discretion.
- Placebo: Placebo matched to ziprasidone capsule orally twice daily up to Week 4.
Period: Overall Study
Arm/Group | Ziprasidone | Placebo
Started | 150 | 88
Treated | 149 | 88
Completed | 97 | 51
Not Completed | 53 | 37
Not completed — Adverse Event | 18 | 13
Not completed — Laboratory abnormality | 1 | 0
Not completed — Lost to Follow-up | 8 | 1
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Other | 16 | 21
Not completed — Randomized, but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Placebo | Total
Number analyzed (Participants) | 149 | 88 | 237
Age, Customized [Number; unit: participants]
  10 to 13 years | 74 | 35 | 109
  14 to 17 years | 74 | 53 | 127
  >=18 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 41 | 106
  Male | 84 | 47 | 131

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Score at Week 4
Description: YMRS: an 11-item scale that measured the severity of manic episodes. Four items were rated on a scale from 0 (symptom absent) to 8 (symptom extremely severe). The remaining items were rated on a scale from 0 (symptom absent) to 4 (symptom extremely severe). YMRS total score ranged from 0 to 60, higher score indicated higher severity of mania.
Time Frame: Baseline, Week 4
Population: Intent-to-treat (ITT): all randomized participants who had baseline measurements, took at least (>=) 1 dose of study medication (ziprasidone or placebo) and had >=1 post-baseline visit. Here, 'n' signifies those participants who were available for this measure at given time points for each group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 143 | 86
units on a scale
  Baseline (n=143,86) | 26.2 (6.6) | 27.0 (6.6)
  Change at Week 4 (n=97,51) | -13.8 (7.8) | -9.9 (7.7)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Change at Week 4: Mixed effects repeated measures Analysis of Covariance (ANCOVA) model with center and participant within center as random effects, treatment, visit and visit-by-treatment interaction as fixed effects and baseline score as a covariate was used for the analysis; Test type: Superiority or Other; p = 0.0005, ANCOVA; Least squares (LS) mean difference = -5.22, 95% CI 2-sided [-8.12 to -2.31], Standard Error of Mean 1.48

2. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Score at Week 1, 2 and 3
Description: as for outcome 1
Time Frame: Baseline, Week 1, 2, 3
Population: ITT population. 'N' (number of participants analyzed) signifies those participants who were available for this measure. 'n' signifies those participants who were available for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 131 | 85
units on a scale
  Change at Week 1 (n=131,85) | -9.3 (7.5) | -6.3 (7.1)
  Change at Week 2 (n=120,81) | -11.5 (8.7) | -8.1 (7.9)
  Change at Week 3 (n=108,65) | -13.0 (8.1) | -9.0 (7.3)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Change at Week 1: Mixed effects repeated measures ANCOVA model with center and participant within center as random effects, treatment, visit and visit-by-treatment interaction as fixed effects and baseline score as a covariate was used for the analysis; Test type: Superiority or Other; p = 0.0006, ANCOVA; LS mean difference = -3.2545, 95% CI 2-sided [-5.1045 to -1.4046], Standard Error of Mean 0.9422
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Change at Week 2: Mixed effects repeated measures ANCOVA model with center and participant within center as random effects, treatment, visit and visit-by-treatment interaction as fixed effects and baseline score as a covariate was used for the analysis; Test type: Superiority or Other; p = 0.0117, ANCOVA; LS mean difference = -3.5857, 95% CI 2-sided [-6.3705 to -0.8009], Standard Error of Mean 1.4184
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; Change at Week 3: Mixed effects repeated measures ANCOVA model with center and participant within center as random effects, treatment, visit and visit-by-treatment interaction as fixed effects and baseline score as a covariate was used for the analysis; Test type: Superiority or Other; p = 0.0047, ANCOVA; LS mean difference = -4.8665, 95% CI 2-sided [-8.2345 to -1.4985], Standard Error of Mean 1.7154

3. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Week 1, 2, 3 and 4
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill).
Time Frame: Baseline, Week 1, 2, 3, 4
Population: ITT population. Here, 'n' signifies those participants who were available for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 143 | 86
units on a scale
  Baseline (n=143,86) | 4.5 (0.7) | 4.5 (0.7)
  Change at Week 1 (n=131,85) | -0.9 (0.8) | -0.5 (0.9)
  Change at Week 2 (n=120,82) | -1.1 (1.0) | -0.6 (0.9)
  Change at Week 3 (n=108,65) | -1.3 (1.0) | -0.7 (1.0)
  Change at Week 4 (n=96,51) | -1.4 (1.1) | -0.9 (0.9)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA; LS mean difference = -0.3754, 95% CI 2-sided [-0.5696 to -0.1812], Standard Error of Mean 0.0989
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS mean difference = -0.5596, 95% CI 2-sided [-0.8256 to -0.2936], Standard Error of Mean 0.1355
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS mean difference = -0.6798, 95% CI 2-sided [-1.0024 to -0.3572], Standard Error of Mean 0.1643
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; Change at Week 4: Mixed effects repeated measures ANCOVA model with center and participant within center as random effects, treatment, visit and visit-by-treatment interaction as fixed effects and baseline score as a covariate was used for the analysis; Test type: Superiority or Other; p = 0.0001, ANCOVA; LS mean difference = -0.6884, 95% CI 2-sided [-1.0342 to -0.3426], Standard Error of Mean 0.1761

4. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale.
Time Frame: Week 1, 2, 3, 4
Population: ITT population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were available for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 132 | 85
units on a scale
  Week 1 (n=132,85) | 2.8 (0.9) | 3.4 (0.9)
  Week 2 (n=120,82) | 2.5 (1.1) | 3.2 (1.1)
  Week 3 (n=108,65) | 2.4 (1.0) | 3.1 (1.3)
  Week 4 (n=96,51) | 2.3 (1.0) | 2.8 (1.1)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 4: Mixed effects repeated measures ANCOVA model with center and participant within center as random effects, treatment, visit and visit-by-treatment interaction as fixed effects was used for the analysis; Test type: Superiority or Other; p = 0.0004, ANCOVA; LS mean difference = -0.76, 95% CI 2-sided [-1.18 to -0.34], Standard Error of Mean 0.21

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Ziprasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 6/149 | 7/88
Other Adverse Events (participants affected / at risk) | 128/149 | 42/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=149) | Placebo (N=88)
Dystonia (Nervous system disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 3
Liver function test abnormal (Investigations) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 2
Hypersexuality (Psychiatric disorders) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=149) | Placebo (N=88)
Vision blurred (Eye disorders) | 9 | 1
Abdominal pain upper (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 21 | 6
Vomiting (Gastrointestinal disorders) | 12 | 1
Fatigue (General disorders) | 23 | 6
Upper respiratory tract infection (Infections and infestations) | 8 | 0
Overdose (Injury, poisoning and procedural complications) | 6 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 8 | 0
Akathisia (Nervous system disorders) | 8 | 1
Dizziness (Nervous system disorders) | 19 | 2
Headache (Nervous system disorders) | 33 | 19
Sedation (Nervous system disorders) | 49 | 5
Somnolence (Nervous system disorders) | 37 | 7
Tremor (Nervous system disorders) | 9 | 0
Insomnia (Psychiatric disorders) | 14 | 3
Restlessness (Psychiatric disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.